CLINICAL TRIAL: NCT05338580
Title: A Multi-center, Open-label Phase II Clinical Trial of TJ271 Injection in Combination With Pembrolizumab in Chinese Patients With Advanced Solid Tumors
Brief Title: Clinical Trial of TJ271 Injection Combined With Pembrolizumab in the Treatment of Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company Development strategy adjustment
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ271001STM202
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: First-line Non-small-cell Lung Cancer; First-line Urothelial Carcinoma; Second-line Urothelial Carcinoma; Second-line Melanoma
Keywords: Evaluate the anti-tumor Efficacy, Safety, Tolerability,Pharmacokinetics and Immunogenicity; A Multi-center, Open-label Phase II Clinical Trial
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TJ271 Injection in Combination with Pembrolizumab (Experimental): TJ271 Injection: 0.9% sodium chloride solution Pembrolizumab: 0.9% sodium chloride solution or 5% glucose solution
  Interventions: Drug: TJ271 Injection in Combination with Pembrolizumab

INTERVENTIONS:
Drug: TJ271 Injection in Combination with Pembrolizumab — TJ271 Injection: 0.9% sodium chloride solution Pembrolizumab: 0.9% sodium chloride solution or 5% glucose solution

SUMMARY:
A Multi-center, Open-label Phase II Clinical Trial of TJ271 Injection in Combination with Pembrolizumab in Chinese Patients with Advanced Solid Tumors to evaluate the anti-tumor efficacy, safety, pharmacokinetics and immunogenicity of TJ271 in combination with pembrolizumab in patients with advanced solid tumors.

DETAILED DESCRIPTION:
A Multi-center, Open-label Phase II Clinical Trial of TJ271 Injection in Combination with Pembrolizumab in Chinese Patients with Advanced Solid Tumors to evaluate the anti-tumor efficacy, safety, pharmacokinetics and immunogenicity of TJ271 in combination with pembrolizumab in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the clinical study; fully understand and sign the written ICF; willing to follow and able to complete all trial procedures.
* Males or females aged => 18 years (inclusive) at the time of signing informed consent.
* With histologically or cytologically confirmed diagnosis of NSCLC, urothelial carcinoma, or melanoma;
* Subjects have at least 1 measurable lesion as defined by RECIST 1.1 (not reside in a field that has been subjected to prior radiotherapy; if within the radiotherapy field, clear evidence of radiographic progression since 14 days after the completion of prior radiotherapy and prior to study enrollment).
* Provide at least 5 unstained tissue sections; with tumor expression levels of PD-L1, CD73, and B7-H3 (central laboratory test) assessed by IHC; the enrollment of NSCLC cohort can be based on the PD-L1 TPS detection level tested by the local laboratory (see 10.5.1.2 Tumor Tissue Sample-Related Biomarkers for details).
* Expected survival => 3 months.
* Main organ function is adequate. See details in the protocol Inclusion Criterion.
* Female subjects of childbearing potential must have a negative urine pregnancy test or serum pregnancy test within 72 hours prior to the first dose of study drug. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Male subjects with reproductive potential and female subjects with pregnancy potential (which refer to men or women who have not been surgically sterilized, and women who are not post-menopausal) must use highly effective contraceptive methods such as oral contraceptives, intrauterine devices, sexual abstinence or barrier contraception in conjunction with spermicides during the course of the study and until 6 months after the last dose.

Exclusion Criteria:

* Diseases amenable to a local curative treatment approach.
* Exclusion criteria for each cohort on prior systemic therapy
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137, B7H3). (Melanoma indications is somewhat special, see inclusion criteria 3.4; if patients received prior CTLA- and discontinued due an irAE, this would be excluded).
* Pregnant or lactating women, or expected to become pregnant or give birth to a child during the study.
* Have received systemic anti-tumor therapy including investigational agents within 4 weeks prior to the start of the study treatment or within five half-lives of the study drug, whichever is shorter.

requiring treatment or hormone replacement may be eligible.

* History of other malignancies within 5 years prior to signing the ICF or other concurrent active malignancies at screening. Patients with localized tumors that have been cured, such as skin basal cell carcinoma, skin squamous cell carcinoma, or cervical carcinoma-in- situ, etc., could be enrolled.
* Has had an allogeneic tissue/solid organ transplant.
* Active autoimmune disease requiring systemic therapy (i.e. use of disease modifying agents, corticosteroids, or immunosuppressive drugs) in past 2 years. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug. (topical, ocular, inhaled or nasal steroids or adrenal replacement therapy of <=10 mg prednisone equivalents is permitted in the absence of active auto-immune disease);
* Currently receiving study treatment in other clinical trials. Subjects who have participated in clinical trials (including trials of investigational vaccines), and received interventional and investigational treatment with invasive and investigational medical devices within 4 weeks prior to the start of the study treatment;
* Subjects who have received major surgeries or experienced severe traumas within 4 weeks prior to the initiation of treatment, or those who are recovering from such surgeries or traumas but the study results will be affected in the opinion of the investigator, or those who have scheduled to undergo surgeries during their participation in the study.
* Therapy to the lung that is >30Gy within 6 months of the first dose of trial treatment. Has received prior radiotherapy within 2 weeks of start of study treatment. or have had a history of radiation pneumonitis.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Hepatitis B:
* Hepatitis C: hepatitis C virus (HCV) antibody positive and meantime HCV RNA [qualitative] is detected.
* Known positive human immunodeficiency virus (HIV) serum reaction.
* With uncontrollable hydrothorax or ascites.
* Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease.
* Clinically significant cardiovascular disease including but not limited to:
* Clinically significant gastrointestinal disorders including:
* Deep vein thrombosis within 6 months prior to the initiation of treatment (except for the case where warfarin has not been used for anti-coagulation for more than 2 weeks prior to treatment initiation).
* Thrombolytic therapy (except for the maintenance of an IV catheter) within 10 days prior to treatment initiation.
* History of uncontrolled seizures within 6 months prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | approximately 2 years
  To evaluate the anti-tumor efficacy of TJ271 in combination with pembrolizumab in patients with advanced solid tumors, i.e. to evaluate the Objective Response Rate (ORR) as per RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided